CLINICAL TRIAL: NCT05390983
Title: Comparison of Carotid Endarterectomy and Repeated Carotid Percutaneous Transluminal Angioplasty With or Without Stenting for In-stent Restenosis
Brief Title: Carotid Endarterectomy vs. Repeated Carotid Angioplasty and Stenting for In-Stent Restenosis
Acronym: CERCAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZ11032017
Record Dates: First submitted 2022-04-19; First posted 2022-05-25 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: In-Stent Carotid Artery Restenosis
Keywords: endarterectomy; percutaneous transluminal angioplasty; stenting; in-stent restenosis
MeSH Terms: interventions — Endarterectomy, Carotid

STUDY DESIGN:
Intervention Model Description: case-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carotid endarterectomy (Experimental): carotid endarterectomy with stent removal
  Interventions: Procedure: Carotid endarterectomy with stent removal
- repeated angioplasty and stenting (Active Comparator): percutaneous transluminal angioplasty with or without stenting
  Interventions: Procedure: Carotid endarterectomy with stent removal

INTERVENTIONS:
Procedure: Carotid endarterectomy with stent removal — Standard carotid endarterectomy will be extended with the stent removal
  Other Names: Carotid endarterectomy

SUMMARY:
Patients with in-stent restenosis in carotid artery indicated to carotid intervention will be randomized into repeated carotid percutaneous transluminal angioplasty with or without stenting or carotid endarterectomy with stent removal. The objective of the randomized study is to compare the safety and effectiveness of CEA and CAS in patients with in-stent restenosis of the ICA.

DETAILED DESCRIPTION:
Patients: Patients with in-stent restenosis in carotid artery indicated to carotid intervention will be randomized into repeated carotid percutaneous transluminal angioplasty with or without stenting or carotid endarterectomy with stent removal.

Repeated carotid percutaneous transluminal angioplasty with or without stenting: Endovascular interventions are going to be performed in local anesthesia from femoral access. Unfractioned heparin (100 IU/kg bodyweight) will be administered in all patients. The procedures will start with diagnostic angiography. Upon verification of severity and morphology of the in-stent stenosis 90 cm long 6F sheath will be introduced into the CCA. The procedures will be performed using distal filter protection. In severe stenoses predilation with 3 or 4 mm diameter balloon will be carried out. In-stent restenoses will be treated preferentially with 5 mm diameter drug eluting balloon. Atropin, up to the dose of 1.0 milligram, can be administered intravenously to prevent serious bradycardia during dilation. Stent will be placed within previous stent in cases of suboptimal PTA result and the decision will be left to the discretion of the interventional specialist. Whenever possible, double-layer technology stent will be used to ensure supreme wall coverage. Distal filter will be removed followed by the completion angiogram including intracranial arteries. Dual antiplatelet therapy (clopidogrel 75 mg/day and acetylsalicylic acid 100 mg/day) will be administered for at least 6 weeks post-procedure. All patients will undergo pre-procedural laboratory testing regarding clopidogrel resistance. In poor responders clopidogrel is going to be replaced by prasugrel or ticagrelor.

Carotid endarterectomy with stent removal: Surgery will be performed in a general or a local anesthesia (decision will be left to the discretion of the operating team) using a cut in front angle of the sternomastoid muscle. Common carotid artery (CCA) and later internal carotid artery (ICA) and external carotid artery (ECA) will be cut free. Common carotid artery, ICA and ECA will be temporarily closed. Using a longitudinal cut of CCA and ICA, stent with an atherosclerotic plaque will be visualized. The stent and a plaque will be withdrawn under the microscopic control and later a suture of arteriotomy will be performed using a monofil non-absorbent fibre 6/0. Just before the end of surgery, hemostatic process will be controlled and drainage will be done. Surgery will be completed by suture of subcutis and cutis. Unfractioned heparin (100 IU/kg bodyweight) could be administered in all patients just before the arteriotomy. In the case of the insufficient collateral flow into middle cerebral artery after clipping of the CCA and ICA, a temporal shunt could be used. Antiplatelet therapy (Aggrenox, clopidogrel 75 mg/day or acetylsalicylic acid 100 mg/day) will be used continuously in all patients.

Clinical examinations: Standard physical and neurologic examinations will be performed before intervention, 24 hours and 30 days after intervention. Evaluation of the neurologic deficit will be performed using the National Institutes of Health Stroke Scale (NIHSS) and modified Rankin scale before, 24 hours and 30 days after intervention.

Randomization: Consecutive patients will be assigned to the carotid endarterctomy with stent removal or repeated carotid percutaneous transluminal angioplasty with or without stenting by a computer-generated 1:1 randomization.

Statistical analysis: All statistical tests will be performed at the Center for Health Research, Faculty of Medicine, University of Ostrava. The normality of distribution of all proceeded data will be checked using the Shapiro-Wilk test. Data with a normal distribution will be reported as the mean ± standard deviation. Parameters not fitting a normal distribution will be presented as the mean, median and interquartile range. Categorical variables in the two arms will be compared by Fisher's exact test. Continuous variables will be compared by the Student's t-test for normally distributed values, or the Mann-Whitney U test. Spearman correlation coefficient and intraclass correlation coefficient will be calculated for the evaluation of interobserver and intraobserver agreements of brain infarction volume measurement. Multiple logistic regression analyses will be used to determine the possible predictors of stroke, TIA, retinal infarction, amaurosis fugax, myocardial infarction or vascular death. All tests will be carried out at an alpha level of significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* In-stent restenosis in carotid artery 70 - 99 %
* Indication to carotid intervention
* Age 18-80 years
* Functionally independent with a modified Rankin score value of 0 - 2 points
* Signed Informed consent

Exclusion Criteria:

* Contraindication to general anesthesia
* Contraindication to angiography (iodine allergy, etc.)
* Technically impossible to perform angioplasty with or without stenting
* Participation in other clinical study within 60 days
* Technically impossible to perform carotid endarterectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
carotid stenosis | 24 hours
  percentage of stenosis in treated carotid artery after intervention

SECONDARY OUTCOMES:
vascular morbidity within 30 days | 30 days
  ischemic stroke, hemorrhagic stroke, myocardial infarction and/or vascular death

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hrbac, MD, PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravskoslezský kraj, Czechia

IPD SHARING:
Plan to Share IPD: No
Data will be available at Mendeley

REFERENCES:
- [Derived] Hrbac T, Fiedler J, Prochazka V, Jonszta T, Roubec M, Pakizer D, Vaclavik D, Netuka D, Heryan T, Skoloudik D. Comparison of carotid endarterectomy and repeated carotid angioplasty and stenting for in-stent restenosis (CERCAS trial): a randomised study. Stroke Vasc Neurol. 2023 Oct;8(5):399-404. doi: 10.1136/svn-2022-002075. Epub 2023 Mar 27. PMID 36972920